CLINICAL TRIAL: NCT06428370
Title: An International Study Investigating the Adoption and Outcome of Damage Control Surgery in Hinchey III-IV Acute Diverticulitis (DACOSAD)
Brief Title: Damage Control Surgery Over the World in Acute Diverticulitis (DACOSAD)
Acronym: DACOSAD
Status: Recruiting | Type: Observational
Sponsor: Link Campus University (Other)
Responsible Party: Sponsor
Other Study IDs: LCU MEDS-06/A 01/2024
Record Dates: First submitted 2024-05-20; First posted 2024-05-24 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-06

CONDITIONS: Diverticular Perforation; Open Abdomen
Keywords: Diverticulitis; Surgery; Open abdomen; Septic shock
MeSH Terms: conditions — Diverticulitis; Shock, Septic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Damage Control Surgery — Simple resection, drop, and open abdomen in case of Hinchey III-IV

SUMMARY:
To analyze the possible benefit of damage control surgery by performing bowel resection, open abdomen, and delayed anastomosis in the treatment of Hinchey III or IV diverticulitis.

DETAILED DESCRIPTION:
Hartmann procedure (HP) is still widely performed in the treatment of purulent or fecal generalized peritonitis as a consequence of a complicated acute large bowel diverticulitis (the so labeled III and IV grade of the Hinchey's classification). More than half of those patients do not undergo to stoma reversal because of its association with significant morbidity and mortality. To date, the use of resection with primary anastomosis (PA) should be preferred, as it is reported in the literature that it is more favorable than HP in terms of morbidity, mortality, and length of postoperative stay. However, PA is often reserved for younger patients with few co-morbidities and a lesser degree of peritoneal contamination while HP is performed in the elderly. Initially described for the treatment of major abdominal injuries, indications for Damage Control Surgery (DCS) have subsequently been extended to septic shock, abdominal compartment syndrome and impossibility to perform a primary closure. In the last decade, DCS has emerged as a valid alternative to HP and Resection-Anastomosis (RA) in patients presenting a severe sepsis caused by purulent or fecal peritonitis in acute diverticulitis. Although DCS is cited as an option in case of impaired hemodynamic status in face of perforated acute diverticulitis, there is still no consensus about such use of DCS. Previous study demonstrated that DCS reduce the Hartmann rate in patients otherwise scheduled for such procedure.

The aim of this study was to describe the potential rationale and outcome of the Damage Control Surgery in patients with purulent and fecal peritonitis.

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 year-old underwent surgery for Hinchey III and IV and submitted to resection, clip and drop, and open abdomen

Exclusion Criteria:

* Subjects <18 year-old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Same as above
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Mortality | 60 days
  Mortality rate related to treatment
Morbidity | 60 days
  Morbidity rate defined by the presence of at least one grade of the Clavien-Dindo Classification scoring system
Total morbidity | 60 days
  Morbidity calculated by means of the Comprehensive Complication Index

SECONDARY OUTCOMES:
Upfront Hartmann rate | 60 days
  Observed to expected (O:E) ratio of Hartmann's procedures
Length of stay (LOS) | 60 days
  Days of stay as inpatient
ICU length of stay | 60 days
  Days of stay in ICU

CONTACTS AND LOCATIONS:
Overall Officials: Gianluca Costa, Prof., Study Director — Link Campus University
Locations (9):
- Hospital de Urgencia Asistencia Publica, Santiago, Chile
- Italy (8):
  - Fondazione Policlinico Universitario Campus Bio-Medico, Rome, Lazio
  - UOC Chirurgia Generale - Ospedale GB Grassi, Ostia Antica, Roma
  - UOC Chirurgia Generale Ospedale Coniugi Bernardini, Palestrina, Roma
  - UOC Chirurgia Generale Ospedale Sant'Anna e San Sebastiano, Caserta
  - UOC Chirurgia Generale, Urgenza e Trauma Pisa University Hospital, Pisa
  - Fondazione Policlinico Universitario "A.Gemelli", Roma
  - UOC Chirurgia Generale ed Urgenza Ospedale Santo Spirito in Sassia, Roma
  - Dipartimento di Chirurgia AOU Policlinico Umberto I Sapienza Università di Roma, Roma

REFERENCES:
- [Background] Perrone G, Giuffrida M, Abu-Zidan F, Kruger VF, Livrini M, Petracca GL, Rossi G, Tarasconi A, Tian BWCA, Bonati E, Mentz R, Mazzini FN, Campana JP, Gasser E, Kafka-Ritsch R, Felsenreich DM, Dawoud C, Riss S, Gomes CA, Gomes FC, Gonzaga RAT, Canton CAB, Pereira BM, Fraga GP, Zem LG, Cordeiro-Fonseca V, de Mesquita Tauil R, Atanasov B, Belev N, Kovachev N, Melendez LJJ, Dimova A, Dimov S, Zelic Z, Augustin G, Bogdanic B, Moric T, Chouillard E, Bajul M, De Simone B, Panis Y, Esposito F, Notarnicola M, Lauka L, Fabbri A, Hentati H, Fnaiech I, Aurelien V, Bougard M, Roulet M, Demetrashvili Z, Pipia I, Merabishvili G, Bouliaris K, Koukoulis G, Doudakmanis C, Xenaki S, Chrysos E, Kokkinakis S, Vassiliu P, Michalopoulos N, Margaris I, Kechagias A, Avgerinos K, Katunin J, Lostoridis E, Nagorni EA, Pujante A, Mulita F, Maroulis I, Vailas M, Marinis A, Siannis I, Bourbouteli E, Manatakis DK, Tasis N, Acheimastos V, Maria S, Stylianos K, Kuzeridis H, Korkolis D, Fradelos E, Kavalieratos G, Petropoulou T, Polydorou A, Papacostantinou I, Triantafyllou T, Kimpizi D, Theodorou D, Toutouzas K, Chamzin A, Frountzas M, Schizas D, Karavokyros I, Syllaios A, Charalabopoulos A, Boura M, Baili E, Ioannidis O, Loutzidou L, Anestiadou E, Tsouknidas I, Petrakis G, Polenta E, Bains L, Gupta R, Singh SK, Khanduri A, Bala M, Kedar A, Pisano M, Podda M, Pisanu A, Martines G, Trigiante G, Lantone G, Agrusa A, Di Buono G, Buscemi S, Veroux M, Gioco R, Veroux G, Oragano L, Zonta S, Lovisetto F, Feo CV, Pesce A, Fabbri N, Lantone G, Marino F, Perrone F, Vincenti L, Papagni V, Picciariello A, Rossi S, Picardi B, Del Monte SR, Visconti D, Osella G, Petruzzelli L, Pignata G, Andreuccetti J, D'Alessio R, Buonfantino M, Guaitoli E, Spinelli S, Sampietro GM, Corbellini C, Lorusso L, Frontali A, Pezzoli I, Bonomi A, Chierici A, Cotsoglou C, Manca G, Delvecchio A, Musa N, Casati M, Letizia L, Abate E, Ercolani G, D'Acapito F, Solaini L, Guercioni G, Cicconi S, Sasia D, Borghi F, Giraudo G, Sena G, Castaldo P, Cardamone E, Portale G, Zuin M, Spolverato Y, Esposito M, Isernia RM, Di Salvo M, Manunza R, Esposito G, Agus M, Asti ELG, Bernardi DT, Tonucci TP, Luppi D, Casadei M, Bonilauri S, Pezzolla A, Panebianco A, Laforgia R, De Luca M, Zese M, Parini D, Jovine E, De Sario G, Lombardi R, Aprea G, Palomba G, Capuano M, Argenio G, Orio G, Armellino MF, Troian M, Guerra M, Nagliati C, Biloslavo A, Germani P, Aizza G, Monsellato I, Chahrour AC, Anania G, Bombardini C, Bagolini F, Sganga G, Fransvea P, Bianchi V, Boati P, Ferrara F, Palmieri F, Cianci P, Gattulli D, Restini E, Cillara N, Cannavera A, Nita GE, Sarnari J, Roscio F, Clerici F, Scandroglio I, Berti S, Cadeo A, Filippelli A, Conti L, Grassi C, Cattaneo GM, Pighin M, Papis D, Gambino G, Bertino V, Schifano D, Prando D, Fogato L, Cavallo F, Ansaloni L, Picheo R, Pontarolo N, Depalma N, Spampinato M, D'Ugo S, Lepre L, Capponi MG, Campa RD, Sarro G, Dinuzzi VP, Olmi S, Uccelli M, Ferrari D, Inama M, Moretto G, Fontana M, Favi F, Picariello E, Rampini A, Barberis A, Azzinnaro A, Oliva A, Totaro L, Benzoni I, Ranieri V, Capolupo GT, Carannante F, Caricato M, Ronconi M, Casiraghi S, Casole G, Pantalone D, Alemanno G, Scheiterle M, Ceresoli M, Cereda M, Fumagalli C, Zanzi F, Bolzon S, Guerra E, Lecchi F, Cellerino P, Ardito A, Scaramuzzo R, Balla A, Lepiane P, Tartaglia N, Ambrosi A, Pavone G, Palini GM, Veneroni S, Garulli G, Ricci C, Torre B, Russo IS, Rottoli M, Tanzanu M, Belvedere A, Milone M, Manigrasso M, De Palma GD, Piccoli M, Pattacini GC, Magnone S, Bertoli P, Pisano M, Massucco P, Palisi M, Luzzi AP, Fleres F, Clarizia G, Spolini A, Kobe Y, Toma T, Shimamura F, Parker R, Ranketi S, Mitei M, Svagzdys S, Pauzas H, Zilinskas J, Poskus T, Kryzauskas M, Jakubauskas M, Zakaria AD, Zakaria Z, Wong MP, Jusoh AC, Zakaria MN, Cruz DR, Elizalde ABR, Reynaud AB, Hernandez EEL, Monroy JMVP, Hinojosa-Ugarte D, Quiodettis M, Du Bois ME, Latorraca J, Major P, Pedziwiatr M, Pisarska-Adamczyk M, Waledziak M, Kwiatkowski A, Czyzykowski L, da Costa SD, Pereira B, Ferreira ARO, Almeida F, Rocha R, Carneiro C, Perez DP, Carvas J, Rocha C, Ferreira C, Marques R, Fernandes U, Leao P, Goulart A, Pereira RG, Patrocinio SDD, de Mendonca NGG, Manso MIC, Morais HMC, Cardoso PS, Calu V, Miron A, Toma EA, Gachabayov M, Abdullaev A, Litvin A, Nechay T, Tyagunov A, Yuldashev A, Bradley A, Wilson M, Panyko A, Lateckova Z, Lacko V, Lesko D, Soltes M, Radonak J, Turrado-Rodriguez V, Termes-Serra R, Morales-Sevillano X, Lapolla P, Mingoli A, Brachini G, Degiuli M, Sofia S, Reddavid R, de Manzoni Garberini A, Buffone A, Del Pozo EP, Aparicio-Sanchez D, Dos Barbeito S, Estaire-Gomez M, Viton-Herrero R, de Los Angeles Gil Olarte-Marquez M, Gil-Martinez J, Alconchel F, Nicolas-Lopez T, Rahy-Martin AC, Pelloni M, Banolas-Suarez R, Mendoza-Moreno F, Nisa FG, Diez-Alonso M, Rodas MEV, Agundez MC, Andres MIP, Moreira CCL, Perez AL, Ponce IA, Gonzalez-Castillo AM, Membrilla-Fernandez E, Salvans S, Serradilla-Martin M, Pardo PS, Rivera-Alonso D, Dziakova J, Huguet JM, Valle NP, Ruiz EC, Valcarcel CR, Moreno CR, Salazar YTM, Garcia JJR, Mico SS, Lopez JR, Farre SP, Gomez MS, Petit NM, Titos-Garcia A, Aranda-Narvaez JM, Romacho-Lopez L, Sanchez-Guillen L, Aranaz-Ostariz V, Bosch-Ramirez M, Martinez-Perez A, Martinez-Lopez E, Sebastian-Tomas JC, Jimenez-Riera G, Jimenez-Vega J, Cuellar JAN, Campos-Serra A, Munoz-Campana A, Gracia-Roman R, Alegre JM, Pinto FL, O'Sullivan SN, Antona FB, Jimenez BM, Lopez-Sanchez J, Carmona ZG, Fernandez RT, Sierra IB, de Leon LRG, Moreno VP, Iglesias E, Cumplido PL, Bravo AA, Simo IR, Dominguez CL, Caamano AG, Lozano RC, Martinez MD, Torres AN, de Quiros JTMB, Pellino G, Cloquell MM, Moller EG, Jalal-Eldin S, Abdoun AK, Hamid HKS, Lohsiriwat V, Mongkhonsupphawan A, Baraket O, Ayed K, Abbassi I, Ali AB, Ammar H, Kchaou A, Tlili A, Zribi I, Colak E, Polat S, Koylu ZA, Guner A, Usta MA, Reis ME, Mantoglu B, Gonullu E, Akin E, Altintoprak F, Bayhan Z, Firat N, Isik A, Memis U, Bayrak M, Altintas Y, Kara Y, Bozkurt MA, Kocatas A, Das K, Seker A, Ozer N, Atici SD, Tuncer K, Kaya T, Ozkan Z, Ilhan O, Agackiran I, Uzunoglu MY, Demirbas E, Altinel Y, Meric S, Hacim NA, Uymaz DS, Omarov N, Balik E, Tebala GD, Khalil H, Rana M, Khan M, Florence C, Swaminathan C, Leo CA, Liasis L, Watfah J, Trostchansky I, Delgado E, Pontillo M, Latifi R, Coimbra R, Edwards S, Lopez A, Velmahos G, Dorken A, Gebran A, Palmer A, Oury J, Bardes JM, Seng SS, Coffua LS, Ratnasekera A, Egodage T, Echeverria-Rosario K, Armento I, Napolitano LM, Sangji NF, Hemmila M, Quick JA, Austin TR, Hyman TS, Curtiss W, McClure A, Cairl N, Biffl WL, Truong HP, Schaffer K, Reames S, Banchini F, Capelli P, Coccolini F, Sartelli M, Bravi F, Vallicelli C, Agnoletti V, Baiocchi GL, Catena F. Goodbye Hartmann trial: a prospective, international, multicenter, observational study on the current use of a surgical procedure developed a century ago. World J Emerg Surg. 2024 Apr 16;19(1):14. doi: 10.1186/s13017-024-00543-w. PMID 38627831
- [Background] Cirocchi R, Sapienza P, Anania G, Binda GA, Avenia S, di Saverio S, Tebala GD, Zago M, Donini A, Mingoli A, Nascimbeni R. State-of-the-art surgery for sigmoid diverticulitis. Langenbecks Arch Surg. 2022 Feb;407(1):1-14. doi: 10.1007/s00423-021-02288-5. Epub 2021 Sep 23. PMID 34557938
- [Background] Sohn M, Agha A, Iesalnieks I, Gundling F, Presl J, Hochrein A, Tartaglia D, Brillantino A, Perathoner A, Pratschke J, Aigner F, Ritschl P. Damage control strategy in perforated diverticulitis with generalized peritonitis. BMC Surg. 2021 Mar 16;21(1):135. doi: 10.1186/s12893-021-01130-5. PMID 33726727
- [Background] Zizzo M, Castro Ruiz C, Zanelli M, Bassi MC, Sanguedolce F, Ascani S, Annessi V. Damage control surgery for the treatment of perforated acute colonic diverticulitis: A systematic review. Medicine (Baltimore). 2020 Nov 25;99(48):e23323. doi: 10.1097/MD.0000000000023323. PMID 33235095
- [Background] Khan A, Hsee L, Mathur S, Civil I. Damage-control laparotomy in nontrauma patients: review of indications and outcomes. J Trauma Acute Care Surg. 2013 Sep;75(3):365-8. doi: 10.1097/TA.0b013e31829cb65e. PMID 23928745
- [Result] Pavlidis ET, Pavlidis TE. Current Aspects on the Management of Perforated Acute Diverticulitis: A Narrative Review. Cureus. 2022 Aug 26;14(8):e28446. doi: 10.7759/cureus.28446. eCollection 2022 Aug. PMID 36176861
- [Result] Tartaglia D, Costa G, Camillo A, Castriconi M, Andreano M, Lanza M, Fransvea P, Ruscelli P, Rimini M, Galatioto C, Chiarugi M. Damage control surgery for perforated diverticulitis with diffuse peritonitis: saves lives and reduces ostomy. World J Emerg Surg. 2019 Apr 16;14:19. doi: 10.1186/s13017-019-0238-1. eCollection 2019. PMID 31015859
- [Result] Berg A, Rosenzweig M, Kuo YH, Onayemi A, Mohidul S, Moen M, Sciarretta J, Davis JM, Ahmed N. The results of rapid source control laparotomy or open abdomen for acute diverticulitis. Langenbecks Arch Surg. 2022 Feb;407(1):259-265. doi: 10.1007/s00423-021-02304-8. Epub 2021 Aug 28. PMID 34455491
- [Result] Costa G, La Torre M, Frezza B, Fransvea P, Tomassini F, Ziparo V, Balducci G. Changes in the surgical approach to colonic emergencies during a 15-year period. Dig Surg. 2014;31(3):197-203. doi: 10.1159/000365254. Epub 2014 Aug 28. PMID 25170867
- [Result] Horesh N, Lessing Y, Rudnicki Y, Kent I, Kammar H, Ben-Yaacov A, Dreznik Y, Avital S, Mavor E, Wasserberg N, Kashtan H, Klausner J, Gutman M, Zmora O, Tulchinsky H. Comparison between laparoscopic and open Hartmann's reversal: results of a decade-long multicenter retrospective study. Surg Endosc. 2018 Dec;32(12):4780-4787. doi: 10.1007/s00464-018-6227-8. Epub 2018 May 15. PMID 29766303
- [Result] Horesh N, Lessing Y, Rudnicki Y, Kent I, Kammar H, Ben-Yaacov A, Dreznik Y, Tulchinsky H, Avital S, Mavor E, Wasserberg N, Kashtan H, Klausner JM, Gutman M, Zmora O. Considerations for Hartmann's reversal and Hartmann's reversal outcomes-a multicenter study. Int J Colorectal Dis. 2017 Nov;32(11):1577-1582. doi: 10.1007/s00384-017-2897-2. Epub 2017 Sep 6. PMID 28879552